CLINICAL TRIAL: NCT02667366
Title: Improving Access to Evidence-based Treatment for Depression: Effectiveness and Cost-effectiveness of Telephone-delivered Cognitive Behavioral Therapy (CBT) in Primary Care
Brief Title: Effectiveness and Cost-effectiveness of Telephone-delivered Psychotherapy for Depression in Primary Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Zurich (Other)
Collaborators: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BW-0417
Record Dates: First submitted 2015-12-03; First posted 2016-01-28 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Depression
Keywords: mild and moderate depression
MeSH Terms: conditions — Depression; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tel-PT (Experimental): Tel-PT receives a manualized short-term CBT. Treatment consists of one initial face-to-face appointment and 8-12 subsequent telephone sessions between patient and licensed therapist. Each telephone contact lasts between 20 and 30 minutes and take place on a weekly and later biweekly basis.
  Interventions: Behavioral: Tel-PT
- TAU and text messages (Active Comparator): Control Group receives treatment as usual and additionally weekly text messages containing general information about depression.
  Interventions: Behavioral: TAU and text messages

INTERVENTIONS:
Behavioral: Tel-PT
  Arms: Tel-PT
Behavioral: TAU and text messages
  Arms: TAU and text messages

SUMMARY:
The aim of the study is the examination of effectiveness and cost-effectiveness of a telephone-based psychotherapy (Tel-PT) for depression compared to treatment as usual in primary care.

DETAILED DESCRIPTION:
The overall purpose of the study is to examine the effectiveness of telephone psychotherapy (Tel-PT) for the treatment of mild to moderate depression on different outcome-levels and under clinically representative conditions in Swiss primary health care. The randomized-controlled trial (RCT) will evaluate the primary hypothesis that Tel-PT is more effective than routine primary care (i.e. treatment as usual, TAU), more specifically, that it leads to significant higher reduction in depression severity than TAU at follow-up.

The intervention group (IG) receives a manualized short-term cognitive behavioral treatment, which is the adapted German version of the program "Creating a balance" developed in the USA. The therapy consists of one face-to-face and 8-12 telephone contacts and is carried out by a licensed psychotherapist.

More concrete, recruitment and inclusion of the patients will be carried out by the participating general practitioners (GPs). GPs will be instructed to screen patients at risk for depression, especially those revealing diffuse somatic symptoms and suffering from chronic diseases. If positively screened, patient's depressive symptoms are assessed with Patient Health Questionnaire (PHQ-9) and diagnosed according to ICD-10.

All GPs will receive an initial training prior to their participation, providing them with study information and procedures as well as training in screening procedure, psychodiagnostics and study enrolment.

Eligible patients are provided with detailed study information and asked to participate. Subsequently, patients will give informed consent. Patients will then be included into the study and fill out the baseline questionnaires (t0). After that, randomization will be carried out at the University of Zurich, based on an appropriately created computer algorithm. Both GPs and patients are informed about the results by the study team within two days. Subsequently, patients in control group (CG) will receive regular text messages and patients in the intervention group (IG) will be called by the study therapist to schedule an initial appointment.

In case of positive results, the overarching objective is the optimization of mental health services for depressed patients by implementing an evidence-based, accessible and cost-effective treatment option into primary care.

ELIGIBILITY:
Inclusion Criteria:

* PHQ-9 score of > 5 and ≤15.
* Informed Consent as documented by signature (Appendix Informed Consent Form)
* Minimum age of 18 years
* Diagnosis of mild to moderate depression according to ICD-10 (F32.0, F32.1, F33.0, F33.1)

Exclusion Criteria:

* Patients currently being in psychotherapeutic treatment or treatment in past three months
* Suicidal tendencies or suicidality
* Insufficient knowledge of German language
* Health condition that does not allow questionnaire completion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-01; Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Change in depressive symptoms | t0 (baseline) and t2 (12 months after baseline)
  The change in depressive symptoms will be assessed with the German version of Patient Health Questionnaire (PHQ-9; Löwe, Spitzer, Zipfel, & Herzog 2002).

SECONDARY OUTCOMES:
Change in depressive symptoms | t0 (baseline) and t1 (four months after baseline)
  The change in depressive symptoms will be assessed with the German version of Patient Health Questionnaire (PHQ-9; Löwe, Spitzer, Zipfel, & Herzog 2002).
Response | t0 (baseline), t1 (four months after baseline), t2 (12 months after baseline)
  Response defined as 50% reduction in the PHQ-9.
Change in health-related quality of life | t0 (baseline), t1 (four months after baseline), t2 (12 months after baseline)
  Change in health-related quality of life is measured with the 12-Item Short Form Health Survey (SF-12; Bullinger & Kirchberger, 1998).
Self-efficacy for management and relapse prevention in depression | t0 (baseline), t1 (four months after baseline), t2 (12 months after baseline)
  Depression self-efficacy scale for management and relapse prevention (Bush et al., 2001).
Cost-effectiveness | t0 (baseline), t1 (four months after baseline), t2 (12 months after baseline)
  Health care utilization and productivity loss will be measured with an adapted version of the Client Sociodemographic and Service Receipt Inventory (CSSRI; Chisholm et al., 2000). For Switzerland, country-specific unit costs will be employed to calculate direct and indirect costs.
Cost-effectiveness | t0 (baseline), t1 (four months after baseline), t2 (12 months after baseline)
  Health-related quality of life for the economic analyses will be measured using the EQ-5D-5L (The EuroQuol Group, 1990), Quality-adjusted life years (QALYs) based on the EQ-5D index will be determined and the incremental cost-effectiveness ratio (ICER) will be computed.

OTHER OUTCOMES:
Acceptance and satisfaction with the intervention | t1 (four months after baseline)
  Patients' and therapists' acceptance and satisfaction with the intervention will be assessed by a self-constructed questionnaire.
Process and structural variable | t1 (four months after baseline), t2 (12 months after baseline)
  Mean duration of telephone contacts
Process and structural variable | t1 (four months after baseline), t2 (12 months after baseline)
  Mean number of telephone contacts.
Process and structural variable | t1 (four months after baseline), t2 (12 months after baseline)
  Dropout rate

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Watzke, Prof, Principal Investigator — University of Zurich, Department of Clinical Psychology and Psychotherapy Research
Locations (1):
- University of Zurich, Zurich, Switzerland

REFERENCES:
- [Background] Löwe, B, Spitzer, RL, Zipfel, S, & Herzog, W. Gesundheitsfragebogen für Patienten (PHQ-D): Manual und Testunterlagen. Pfizer. Karlsruhe: 2002.
- [Background] Watzke B, Heddaeus D, Steinmann M, Konig HH, Wegscheider K, Schulz H, Harter M. Effectiveness and cost-effectiveness of a guideline-based stepped care model for patients with depression: study protocol of a cluster-randomized controlled trial in routine care. BMC Psychiatry. 2014 Aug 20;14:230. doi: 10.1186/s12888-014-0230-y. PMID 25182269
- [Background] Simon GE, Ludman EJ, Tutty S, Operskalski B, Von Korff M. Telephone psychotherapy and telephone care management for primary care patients starting antidepressant treatment: a randomized controlled trial. JAMA. 2004 Aug 25;292(8):935-42. doi: 10.1001/jama.292.8.935. PMID 15328325
- [Background] Bush, T, Russo, J, Ludman, E, Lin, E, Von Korff, M, Simon, G, Walker, E. Perceived self-efficacy for depression self-management. A reliable and valid self-report measure with predictive validity: Poster presentation at the American Psychological Society Meeting, June 2001. Toronto, Canada.
- [Background] Bullinger, M, & Kirchberger, I. Fragebogen zum Gesundheitszustand. Hogrefe. Göttingen: 1998.
- [Derived] Haller E, Besson N, Watzke B. "Unrigging the support wheels" - A qualitative study on patients' experiences with and perspectives on low-intensity CBT. BMC Health Serv Res. 2019 Oct 9;19(1):686. doi: 10.1186/s12913-019-4495-1. PMID 31597555
- [Derived] Watzke B, Haller E, Steinmann M, Heddaeus D, Harter M, Konig HH, Wegscheider K, Rosemann T. Effectiveness and cost-effectiveness of telephone-based cognitive-behavioural therapy in primary care: study protocol of TIDe - telephone intervention for depression. BMC Psychiatry. 2017 Jul 19;17(1):263. doi: 10.1186/s12888-017-1429-5. PMID 28724423